CLINICAL TRIAL: NCT05365165
Title: Researching the Affect of Sevoflurane Application for Maintenance of Anesthesia During Aortic Cross-clamping in Cardiac Surgery on Delirium
Brief Title: Researching the Affect of Sevoflurane in Cardiac Surgery on Delirium
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Aysegul Cigdem Caglayan, MD, Anesthesiology and Reanimation, Derince Training and Research Hospital
Other Study IDs: DERINCETRHCCAGLAYAN002
Record Dates: First submitted 2022-04-24; First posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium | interventions — Sevoflurane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- sevoflurane: Standard anesthesia management will be applied in the induction and maintenance of anesthesia. In the induction of anesthesia 1mg/kg lidocaine , 1.5-2mg/kg propofol , 1 mcg /kg fentanyl citrate, 0.6 mg/kg rocuronium bromide will be administered. Sevoflurane for maintenance of anesthesia and propofol and fentanyl if needed bolus will be applied. BIS monitoring will be performed to control the depth of anesthesia.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane — Sevoflurane will be applied during aortic cross- clamping in cardiac surgery

SUMMARY:
Many risk factors have been identified for delirium after open heart surgery . One of the main risk factors; duration of stay on mechanical ventilator . Our hypothesis; The use of sevoflurane during aortic cross-clamping reduces the need for long-acting intravenous anesthetic agents. Therefore, patients will be weaned from the mechanical ventilator in a shorter time. Patients with shorter stays on mechanical ventilation develop less postoperative delirium.

DETAILED DESCRIPTION:
Standard anesthesia management will be applied in the induction and maintenance of anesthesia. In the induction of anesthesia 1mg/kg lidocaine , 1.5-2mg/kg propofol , 1 mcg /kg fentanyl citrate, 0.6 mg/kg rocuronium bromide will be administered. Sevoflurane for maintenance of anesthesia and propofol and fentanyl if needed bolus will be applied. BIS monitoring will be performed to control the depth of anesthesia. Patients' peroperative hemodynamic levels, arterial blood gas levels, operation time, pump time, aortic cross clamp time, postoperative complications , the amount of blood and fluid used, the amount of iv anesthetic used, the extubation time, the length of stay in the intensive care unit, the length of stay in the hospital will be followed and recorded. Postoperative delirium follow-ups of the patients will be recorded once a day by the same investigator using the Nursing Delirium Screening Scale and Delirium Rating Scale Revised-98 until they are discharged from the hospital .

ELIGIBILITY:
Inclusion Criteria:

Patients with a score of 25 and above in the mini-mental state test performed in the preoperative period

Exclusion Criteria:

Those who are scheduled for emergency surgery

Those with known dementia and/or neurological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who will have elective open heart surgery, patients over the age of 18, and patients with a score of 25 and above in the mini mental state test performed in the preoperative period will be included in the study.
Sampling Method: Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
rate of delirium after open heart surgery | up to 2 weeks
  Postoperative delirium follow-ups of the patients will be recorded once a day by the same investigator using the Nursing Delirium Screening Scale and Delirium Rating Scale Revised-98 until they are discharged from the hospital. The Nu-DESC is a 5-item observation scale that can be completed quickly. Each item is evaluated on a 3-point Likert (from 0 to 3). The total score is obtained by adding the values of the items, and the highest score is 10. If the total score is 2 and above, the diagnosed of delirium is made. The DRS-R-98 is a 16-item scale with a maximum total scale score of 46 points and a maximum severity score of 39 points. A suggested cut-off score for delirium is >19 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Ayşegül Çiğdem Çağlayan, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided